CLINICAL TRIAL: NCT04159506
Title: Feasibility and Acceptability of The Equus Effect: A Small Randomized Controlled Pilot Study of an Equine-facilitated Therapy
Brief Title: Feasibility and Acceptability Off The Equus Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3312-P; 02342-003 (Other Grant/Funding Number: VA Connecticut Healthcare System)
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Social Skills; Emotional Dysfunction
Keywords: equine therapy; social functioning; emotion regulation
MeSH Terms: conditions — Social Skills; Social Adjustment; Emotional Regulation | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized to receive either 1) The Equus Effect (TEE) or 2) attention control (AC), both group interventions. Each week, the 4-session TEE will include 1) mindfulness activities, 2) emotion regulation and interpersonal skills education, 3) experiential activities with horses incorporating opportunities to develop emotion regulation and interpersonal skills, and 4) between-session application of lessons learned from the equine activities. AC will have similar elements without equine features.
Who Masked: Outcomes Assessor
Masking Description: The research assistant who will collect study assessments will not know the randomization of participants to conditions. Randomization will be conducted by the study coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Equus Effect (TEE) (Experimental): TEE is a 4-session intervention. Each session is 4 hours and includes: 1) mindfulness-based activities; 2) didactics about emotion regulation and interpersonal skills; and 3) experiential learning activities with horses that provide opportunities to practice emotion regulation and interpersonal skills. At the end of each session, Veterans debrief about what they learned and identify how they might apply this knowledge to manage their mental health concerns and function better socially.
  Interventions: Behavioral: mindfulness, emotion didactics, interpersonal skills, experiential learning
- Attention Control (AC) (Active Comparator): AC will exclude equine-related activities or discussions but maintain mindfulness-based activities, emotion regulation and interpersonal skills didactics, and experiential learning activities with between-session application. Instead of experiential equine activities, AC will rely on team-building activities, which aim to enhance social relations by involving participants in collaborative tasks and providing opportunities for emotion regulation and interpersonal skills practice.
  Interventions: Behavioral: mindfulness, emotion didactics, interpersonal skills, experiential learning

INTERVENTIONS:
Behavioral: mindfulness, emotion didactics, interpersonal skills, experiential learning — mindfulness interventions involve body scanning, deep breathing, and muscle relaxation. Emotion didactics focus on emotion recognition and regulation. Interpersonal skill development looks at how to use emotion regulation to improve social functioning. Experiential learning means learning either through interactions with horses or via team-building activities.

SUMMARY:
The VA Office of Patient Centered Care and Cultural Transformation's Whole Health initiative promotes the use of complementary and integrative health (CIH) approaches with traditional medical care to help Veterans achieve meaningful life goals and improved functioning. Equine-facilitated therapy (EFT), an animal-assisted form of CIH, is increasingly available to Veterans within the VA. Horses have extreme sensitivity to the emotional states, behaviors, and intentions of their herds and other animals, including humans, and mirror body language and respond to subtle nonverbal cues. As such, horses have the capacity to provide immediate feedback about a people's emotional and behavioral states. This capacity affords people opportunities to become more emotionally self-aware and, with guidance from EFT facilitators, learn how to regulate emotions and become calmer and more patient, attentive, and confident to gain the horses' cooperation. Participants in EFT are encouraged to apply what they have learned from their equine experiences to their relationships with people. Since high quality social functioning depends on effective regulation of one's emotions, EFT offers a novel way in which to improve the social functioning of Veterans with mental health concerns. VAs are increasingly embracing EFT as a CIH. However, carefully conducted, scientifically valid research about EFT has not been conducted. Existing peer-reviewed research about EFT for mental health is very limited, of poor methodological quality, and not focused on adults. None of it targets social functioning as a main outcome. This small randomized controlled pilot study proposes to examine an innovative EFT called The Equus Effect (TEE) as a complement to Veterans' existing VA mental health services to improve social functioning. TEE aims to improve Veterans' social functioning by developing their emotion regulation and interpersonal skills through therapeutic interactions with horses. This study will evaluate 1) the feasibility of study procedures, assessments, and outcomes, 2) the fidelity of experimental and control interventions, and 3) the acceptability of the interventions to Veterans and their mental health clinicians using mixed quantitative-qualitative methods. The study has the potential to lend initial credibility to the therapeutic claims of this increasingly popular CIH.

DETAILED DESCRIPTION:
**Please note that as a consequence of the COVID-19 pandemic, and after consultation with the appropriate research oversight, regulatory and monitoring entities, screening and enrollment was placed on temporary administrative hold from 04/30/2020 - 3/31/2022. Experimental and comparator conditions had to occur in person, in groups, and with van transportation to and from the intervention site. The study resumed preparations for the pilot trial 4/1/2022 and began participant screening and recruitment 6/15/2022.**

The VA Office of Patient Centered Care and Cultural Transformation launched the Whole Health initiative to transform the Veterans Health Administration into a healthcare system in which providers and Veterans develop holistic, personalized, proactive, patient-driven healthcare plans that center on realizing meaningful life goals and improved functioning. Whole Health promotes the use of complementary and integrative health (CIH) approaches with traditional medical care to achieve these aims - consistent with psychosocial rehabilitation's emphasis on recovery-oriented, community-based functional outcomes. Equine-facilitated therapy (EFT), an animal-assisted form of CIH, is increasingly available to Veterans within the VA. Horses are prey animals with extreme sensitivity to the emotional states, behaviors, and intentions of their herds and other animals, including humans, and mirror body language and respond to subtle nonverbal cues. As such, horses have the capacity to provide immediate feedback about a person's emotional and behavioral states (e.g., pinning ears back when someone is angry or relaxing them forward when a person is calm). As a person interacts with horses, this capacity affords him or her an opportunity to become more emotionally self-aware and, with guidance from EFT facilitators, learn how to regulate emotions and become calmer and more patient, attentive, and confident to gain the horses' cooperation. With EFT, emotion regulation is the key mechanism for social interaction with horses, and participants in EFT are encouraged to apply what they have learned from their equine experiences to their relationships with people. Since high quality social functioning depends on effective regulation of one's emotions, EFT offers a novel way in which to improve the social functioning of Veterans with mental health concerns. In fact, in the VA, EFT has been used to address a variety of diagnostic issues commonly experience by Veterans, including PTSD, depression, anxiety, substance use and eating disorders. However, peer-reviewed published quantitative and qualitative research on EFT as a CIH for mental health is very limited, of poor methodological quality, and focused on school-age children and adolescents, not adults. None of it targets social functioning as a main outcome. Given VAs increasing embrace of EFT as a CIH, carefully conducted research that aims to systematically develop and study EFT for Veterans is sorely needed to ensure that EFT is feasible to study, acceptable to Veterans and clinicians, and clinically promising.

The investigators propose to pilot test an innovative EFT called The Equus Effect (TEE) as a complement to Veterans' existing VA mental health services to improve social functioning. TEE aims to improve Veterans' social functioning by developing their emotion regulation and interpersonal skills through therapeutic interactions with horses. In line with recommendations for pilot investigations, the investigators will conduct a randomized pilot study to 1) evaluate the feasibility of study procedures, assessments, and outcomes, 2) demonstrate experimental and control interventions can be delivered with fidelity, and 3) examine the acceptability of the interventions. To accomplish these goals, the investigators will enroll a transdiagnostic cohort of 40 Veterans involved in VA mental health services with social dysfunction and emotion dysregulation. Participants will be randomized to receive either 1) TEE or 2) attention control (AC), both group interventions. Each week, the 4-session TEE will include 1) mindfulness activities, 2) emotion regulation and interpersonal skills education, 3) experiential activities with horses incorporating opportunities to develop emotion regulation and interpersonal skills, and 4) between-session application of lessons learned from the equine activities. AC will have similar elements without equine features. Intervention outcomes will be measured at 4- and 16-weeks post randomization. Specifically, using mixed quantitative-qualitative methods, the investigators aim to:

Aim 1: Determine the feasibility of recruitment, randomization, retention, assessment procedures, and implementation of TEE and AC. Hypothesis: Rates of recruitment will be at least 8 participants per month, and Veterans randomized to TEE will attend intervention sessions, remain in the study, and experience clinically significant changes in social functioning and emotion dysregulation at rates equal to or superior to AC.

Aim 2: Demonstrate TEE and AC can be delivered with fidelity. Hypothesis: Facilitators will deliver each intervention consistently and as intended across sessions.

Aim 3: Establish acceptability of TEE and AC by assessing intervention credibility and satisfaction and the usefulness of TEE as a complementary mental health intervention using mixed quantitative-qualitative methods. Hypothesis: Veterans will find TEE and AC credible and satisfying and Veterans and their mental health clinicians will qualitatively report the therapeutic benefits of TEE as a CIH for mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

* seeing a VA Connecticut mental health clinician at least 3 times in the past 3 months with intent to remain in treatment during study enrollment;
* age 18 and over;
* social dysfunction (score > 2.5 on the Social Adjustment Scale-Self Report (SAS-SR) and > 1.5 on Inventory of Interpersonal Problems-32 (IIP-32);
* emotion dysregulation (score > 95 on the Difficulties in Emotion Regulation Scale (DERS);
* sufficient mobility to participate in study procedures, as determined by PI;
* consent to all study procedures, including audio recording of TEE and AC sessions.

Exclusion Criteria:

* psychotic disorder per self-report and verified in medical record or as determined by the Mini-International Neuropsychiatric Interview (MINI);
* acute suicidality;
* inability to read English or communicate in spoken English;
* anticipated unavailability to the study during the next 20 weeks;
* participation in any equine-facilitated therapy in the past 24 weeks;
* unavailability of a landline or cellular telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Martino, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a small pilot study to determine feasibility and acceptability of testing equine-facilitated therapy within a randomized clinical trial design. It will not establish efficacy of the intervention, per se. Nonetheless, the PI will review and consider requests for sharing data with other investigators, after the PI has fully analyzed and published data generated from this trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After one year of study completion
Access Criteria: Interested parties may email the PI to request data sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2022 and February 2023 veterans were recruited through direct-to-participant advertising involving posting VA Connecticut IRB approved flyers in clinical spaces and research recruitment boards at outpatient mental health clinics, intensive outpatient/rehabilitation programs, and a community care center. Initial phone or in-person contact with potential participants offered study information and invitation to complete a preliminary screener to determine potential study eligibility.
Pre-assignment Details: After the preliminary screener, veterans completed a secondary screening that included completing the Mini-International Neuropsychiatric Interview (MINI) to rule out a psychotic disorder, as well as the Social Adjustment Scale-Self Report (SAS-SR); Inventory of Interpersonal Problems-32 (IIP-32); and Difficulties in Emotion Regulation Scale (DERS) to further determine inclusion and exclusion criteria and ensure minimal threshold levels of social dysfunction and emotion dysregulation.
Period: Overall Study
Arm/Group | The Equus Effect (TEE) | Attention Control (AC)
Started | 16 | 15
Completed | 14 | 10
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- The Equus Effect (TEE): TEE is a 4-session intervention. Each session is 4 hours and includes: 1) mindfulness-based activities; 2) didactics about emotion regulation and interpersonal skills; and 3) experiential learning activities with horses that provide opportunities to practice emotion regulation and interpersonal skills. At the end of each session, Veterans debrief about what they learned and identify how they might apply this knowledge to manage their mental health concerns and function better socially.
  mindfulness, emotion didactics, interpersonal skills, experiential learning: mindfulness interventions involve body scanning, deep breathing, and muscle relaxation. Emotion didactics focus on emotion recognition and regulation. Interpersonal skill development looks at how to use emotion regulation to improve social functioning. Experiential learning means learning either through interactions with horses.
- Attention Control (AC): AC will exclude equine-related activities or discussions but maintain mindfulness-based activities, emotion regulation and interpersonal skills didactics, and experiential learning activities with between-session application. Instead of experiential equine activities, AC will rely on team-building activities, which aim to enhance social relations by involving participants in collaborative tasks and providing opportunities for emotion regulation and interpersonal skills practice.
  mindfulness, emotion didactics, interpersonal skills, experiential learning: mindfulness interventions involve body scanning, deep breathing, and muscle relaxation. Emotion didactics focus on emotion recognition and regulation. Interpersonal skill development looks at how to use emotion regulation to improve social functioning. Experiential learning means learning either through team-building activities.
- Total: Total of all reporting groups
Arm/Group | The Equus Effect (TEE) | Attention Control (AC) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.81 (16.73) | 49.47 (13.65) | 49.65 (15.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 14 | 11 | 25
  Female | 1 | 4 | 5
  Nonbinary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 16 | 10 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 7 | 23
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Social Adjustment Scale-Self Report (SAS-SR)
Description: SAS-SR details social functioning in a range of role areas (e.g., work, social and leisure, family); the overall SAS-SR score is 1 (no impairment), to 5 (highest impairment).
Time Frame: Baseline, 4-weeks post-randomization, 16-weeks post-randomization
Population: Full sample of 31 participants was used in baseline analyses. 26 participants had complete data for 4-week post-randomization. 24 participants had complete data for 16-week post-randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Equus Effect (TEE) | Attention Control (AC)
Number analyzed (Participants) | 16 | 15
score on a scale
  Baseline | 2.92 [2.30 to 3.46] | 2.92 [2.12 to 4.46]
  4-week post-randomization: number analyzed (Participants) | 14 | 12
  4-week post-randomization | 2.30 [1.46 to 3.40] | 2.32 [1.26 to 3.50]
  16-week post-randomization: number analyzed (Participants) | 14 | 10
  16-week post-randomization | 2.56 [1.34 to 2.83] | 2.57 [1.58 to 3.80]
Statistical Analysis 1: Comparison: The Equus Effect (TEE) vs Attention Control (AC); Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — This pilot study was designed mostly to determine feasibility and acceptability of TEE, AC, and study methods. Nonetheless, Paired Difference Signed Rank Tests were used to compare conditions given small sample and non-normal distribution of data; No adjustments were made given this was a pilot study focused on feasibility and acceptability; Median Difference (Final Values) = 0.63

2. Primary Outcome: Inventory of Interpersonal Problems-32 (IIP-32)
Description: IIP-32 taps people's interpersonal difficulties across role areas; the IIP-32 total score is 0 (no difficulties), to 4 (extreme difficulties).
Time Frame: Baseline, 4-weeks post-randomization, 16-weeks post-randomization
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Equus Effect (TEE) | Attention Control (AC)
Number analyzed (Participants) | 16 | 15
score on a scale
  Baseline | 2.06 [1.43 to 3.37] | 1.62 [.50 to 2.81]
  4-week post-randomization: number analyzed (Participants) | 14 | 12
  4-week post-randomization | 1.59 [1.21 to 2.37] | 1.76 [.34 to 2.59]
  16-week post-randomization: number analyzed (Participants) | 14 | 10
  16-week post-randomization | 1.48 [.34 to 2.40] | 1.18 [.43 to 2.93]
Statistical Analysis 1: Comparison: The Equus Effect (TEE) vs Attention Control (AC); This pilot study was designed mostly to determine feasibility and acceptability of TEE, AC, and study methods. Nonetheless, Paired Difference Signed Rank Tests were used to compare conditions given small sample and non-normal distribution of data; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); No adjustments were made given this was a pilot study focused on feasibility and acceptability; Median Difference (Final Values) = 0.31

3. Secondary Outcome: Difficulties in Emotion Regulation Scale (DERS)
Description: DERS scores range from 36-180, with higher scores indicating more emotion dysregulation.
Time Frame: Baseline, 4-weeks post-randomization, 16-weeks post-randomization
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Equus Effect (TEE) | Attention Control (AC)
Number analyzed (Participants) | 16 | 15
score on a scale
  Baseline | 119.00 [95.00 to 170.00] | 113.00 [95.00 to 149.00]
  4-week post-randomization: number analyzed (Participants) | 14 | 12
  4-week post-randomization | 117.00 [48.00 to 154] | 107 [61.00 to 150.00]
  16-week post-randomization: number analyzed (Participants) | 14 | 10
  16-week post-randomization | 114.00 [68.00 to 130.00] | 107.50 [43 to 151]
Statistical Analysis 1: Comparison: The Equus Effect (TEE) vs Attention Control (AC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); No adjustments were made given this was a pilot study focused on feasibility and acceptability; Median Difference (Final Values) = 0.67

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from June 2022 through July 2023, the period of time when all screening, baseline and 4-week and 16-week post-randomization assessments occurred.
Description: clinicaltrials.gov definitions were used.
Arm/Group | The Equus Effect (TEE) | Attention Control (AC)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 0/16 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Equus Effect (TEE) (N=16) | Attention Control (AC) (N=15)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was hospitalized for mental health decompensation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Equus Effect (TEE) (N=16) | Attention Control (AC) (N=15)
suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported suicide ideation when completing the MINI; ideation was passive without intent or plan.

LIMITATIONS AND CAVEATS:
The pilot study had a small sample size not powered to detect statistically significant differences in clinical outcomes. It also examined the feasibility and acceptability of one specific equine-facilitated therapy; other equine-facilitated therapy programs may differ from the one we studied. Finally, follow-up was 3-months post-intervention. The feasibility of studying longer follow-up periods was not examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT04159506/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT04159506/ICF_000.pdf